CLINICAL TRIAL: NCT07200258
Title: Changes in Soft Tissue Thickness Following Multiple Coronally Advanced Tunnel (MCAT) vs Vestibular Incision Subperiosteal Tunnel Access (VISTA): A Randomized Clinical Trial With 3D Volumetric Analysis
Brief Title: Changes in Soft Tissue Thickness Following Multiple Coronally Advanced Tunnel (MCAT) vs Vestibular Incision Subperiosteal Tunnel Access (VISTA)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCM_MCAT-VISTA RCT
Record Dates: First submitted 2025-07-14; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-07

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 : Vestibular Incision Subperiosteal Tunnel Access (VISTA) (Experimental): Patients in this arm will receive the Vestibular Incision Subperiosteal Tunnel Access (VISTA) technique, involving remote vestibular incisions and subperiosteal tunneling to treat multiple gingival recessions. A connective tissue graft (CTG) will be inserted and stabilized using a coronally anchored suturing technique.
  Interventions: Procedure: Vestibular Incision Subperiosteal Tunnel Access (VISTA)
- Arm 2 : Modified Coronally Advanced Tunnel Technique (MCAT) (Experimental)
  Interventions: Procedure: Modified Coronally Advanced Tunnel (MCAT)

INTERVENTIONS:
Procedure: Vestibular Incision Subperiosteal Tunnel Access (VISTA) — Remote incisions will be performed in the test group. The VISTA technique will be performed as described by Zadeh (Zadeh, 2011).
  After administration of local anaesthesia, an access incision will be made in the vestibulum to permit elevation of a broad subperiosteal tunnel. A specialized periosteal elevator will be used to create the tunnel by dissecting beneath the periosteum, extending at least one tooth beyond the recession defects and under each papilla, without surface incisions at the gingival margin. The connective tissue graft will be inserted and positioned beneath the tunnel through the incision. A coronally anchored suturing technique will be used. This technique mean placing a horizontal mattress suture using a 6.0 suture with at approximately 2 to 3 mm apical to the gingival margin of each tooth, covering the width of the tooth. If keratinized gingiva is present, the suture will be placed within the band of keratinized gingiva.
  Arms: Arm 1 : Vestibular Incision Subperiosteal Tunnel Access (VISTA)
Procedure: Modified Coronally Advanced Tunnel (MCAT) — In the MCAT group, the surgical approach will follow the technique described by Aroca et al. (2010). After sulcular incisions made without releasing incisions, a full-thickness muco-periosteal tunnel will be carefully elevated beyond the mucogingival junction and under adjacent papillae using tunneling instruments. The root surfaces will be planed, and a subepithelial connective tissue graft will be harvested from the palatal donor site and inserted into the tunnel. Suspended horizontal mattress sutures will be placed around the contact points to advance and stabilize the flap in a position coronal to the cemento-enamel junction (CEJ) (previous composite at the contact point if necessary). Postoperative care will be identical to that described for the VISTA group.
  Arms: Arm 2 : Modified Coronally Advanced Tunnel Technique (MCAT)

SUMMARY:
This randomized clinical trial will compare two surgical methods for treating multiple adjacent gingival recessions (types RT1 and RT2): the Modified Coronally Advanced Tunnel (MCAT) and the Vestibular Incision Subperiosteal Tunnel Access (VISTA). Both methods will use connective tissue grafts (CTG), which are the best way to cover roots.

The main objective is to use three-dimensional (3D) digital volumetric analysis to look at how the thickness of soft tissue has changed after six and 12 months. Secondary outcomes include root coverage, esthetic outcomes, gingival health parameters, hypersensitivity, patient satisfaction, and wound healing quality.

There will be 44 volunteers, and they will be randomly assigned to one of the two surgical methods. Under the same settings, periodontal specialists in training will undertake the procedures at the Universidad Complutense de Madrid. There will be follow-up evaluations at different times up to 12 months after the procedure. The results of this study will help determine whether remote incisions via the VISTA technique offer improved outcomes compared to the MCAT technique.

DETAILED DESCRIPTION:
Parallel group, clinical evaluator and statistician blinded, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally and systemically healthy adults (age ≥ 18 years).
* At least two adjacent sites exhibiting gingival recessions classified as recession type 1 (RT1) o type 2 (RT2) (Cairo et al., 2011), associated with dental hypersensitivity or aesthetic concerns.
* Presence ≥2 mm depth on at least one recession
* Smokers ≤ 10 cigarettes.
* Full-mouth plaque and bleeding scores ≤20%.
* Patients being able to maintain good oral hygiene.

Exclusion Criteria:

* Compromised general health.
* Pregnancy or attempting to get pregnant (self-reported).
* Untreated periodontal diseases
* Presence of: (i) severe tooth malposition; (ii) root caries or inadequate prosthetic restorations; (iii) previous periodontal plastic surgery at the experimental sites.
* Smokers >10 cigarettes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Areal Marginal Soft Tissue Thickness (aTHK) | Baseline, 3, 6 and 12 months post-surgery
  Soft tissue thickness will be measured using volumetric analysis of STL digital intraoral scans. The region of interest (ROI) corresponds to the previously exposed root surface. The volume difference between baseline and follow-up scans (6 months) will be divided by the surface area leading to an areal thickness (aTHK), expressed in millimeters.

SECONDARY OUTCOMES:
Mean Root coverage | 3, 6 and 12 months
  Percentage of root coverage compared with baseline recession depth. Unit of Measure: % Measurement Tool: UNC-15 periodontal probe
Recession Depth | Baseline, 3 , 6 and 12 months
  Distance from gingival margin to cemento-enamel junction (GM-CEJ). Unit of Measure: mm Measurement Tool: UNC-15 periodontal probe
Probing Pocket Depth | baseline, 3, 6 and 12 months.
  Distance from the gingival margin to the bottom of the sulcus at the mid-buccal site.
  Unit of Measure: mm Measurement Tool: UNC-15 periodontal probe
Keratinized tissue Width | baseline, 3, 6 and 12 months.
  Distance from gingival margin to mucogingival junction.
  Unit of Measure: mm
  Measurement Tool: UNC-15 periodontal probe
Gingival Thickness | baseline, 3, 6 and 12 months.
  Gingival phenotype assessed by probe transparency.
  Unit of Measure: Thick/Thin (categorical)
  Measurement Tool: UNC-15 periodontal probe
Loss of Attachment | Baseline, 3, 6 and 12 months.
  Presence or absence of interproximal clinical attachment loss at treated sites.
  Unit of Measure: mm
  Measurement Tool: UNC-15 periodontal probe
Root Coverage Esthetic Score | 3 6 and 12 months.
  Esthetic evaluation of root coverage outcomes (0-10 composite score).
  Unit of Measure: Score (0-10)
  Measurement Tool: RES index (Cairo 2009) from standardized photographs
Dental Hypersensitivity | baseline, 3, 6 and 12 months
  Sensitivity to air stimulus at cervical area.
  Unit of Measure: Frequency (%) of teeth with sensitivity
  Measurement Tool: Standardized air-blast test (10 seconds)
Flap Tension | Baseline
  Residual flap tension during coronal advancement.
  Unit of Measure: Newtons (N)
  Measurement Tool: Calibrated tension meter (Burkhardt & Lang, 2010)
Oral Health Impact Profile | Baseline, 3 6 and 12 month
  Patient-reported outcomes using the OHIP-14 questionnaire.
  Unit of Measure: Score (0-56; higher = worse QoL)
  Measurement Tool: Validated Spanish version of OHIP-14
Patients Concerns with recession | Baseline, 6 and 12 month
  Patient concerns related to gingival recession will be measured with a condition-specific health-related quality-of-life instrument using a custom 5-point Likert-scale questionnaire assessing five questions: esthetic concern, sensitivity to cold, sensitivity to brushing, root/tooth wear, and fear of tooth loss. Each item is rated from 1 ("not concerned") to 5 ("extremely concerned"). Changes in scores over time will be used to evaluate perceived improvement.
Time to recovery | from baseline to 14 days post surgery
  Number of days until patient-reported recovery after surgery. Recovery is defined as "no or slight trouble" (score 1-2) on all items of the Post-op diary, and pain ≤2 cm on VAS.
  Unit of Measure: Days
  Measurement Tool: Periodontal Surgery Post-op (PS Postop) diary with VAS (0-10 cm) and Likert scales
Digital recession depth | Baseline, 3 6 and 12 month
  Apico-coronal extension of recession measured digitally.
  Unit of Measure: mm
  Measurement Tool: Intraoral scanner (3Shape TRIOS) and Nemotec software
Digital Complete root coverage | Baseline, 3 6 and 12 month
  Whether gingival margin reached/surpassed CEJ.
  Unit of Measure: Binary (Yes/No)
  Measurement Tool: Intraoral scanner (3Shape TRIOS) and Nemotec software
Digital Percentage of root coverage | Baseline, 3 6 and 12 month
  Percentage of root coverage compared with baseline, digitally measured.
  Unit of Measure: %
  Measurement Tool: Intraoral scanner (3Shape TRIOS) and Nemotec software
Digital Pointwise Marginal Soft Tissue Thickness | Baseline, 3 6 and 12 month
  Gingival thickness at specific points in cross-section.
  Unit of Measure: mm
  Measurement Tool: Intraoral scanner (3Shape TRIOS) and Nemotec software
Surgery duration | During Surgery
  Total duration of surgical procedure.
  Unit of Measure: Minutes
  Measurement Tool: Stopwatch (recorded intraoperatively)
Full mouth plaque Score | Baseline 3 6 and 12 months
  Plaque presence will be recorded at six sites per tooth using a periodontal probe and expressed as the percentage of plaque-positive sites over the total number of sites examined.
Full mouth bleeding Score | Baseline, 3 6 and 12 month
  Bleeding on probing will be recorded at six sites per tooth. The FMBS will be calculated as the percentage of sites showing bleeding after probing with a periodontal probe over the total number of sites examined.
Wound Healing Index | Day 7, week 2 , Week 4 and 3 months
  Wound healing will be evaluated using a modified semi-quantitative composite index based on the methodology described by Tonetti (Tonetti et al., 2018).
  Healing is assessed evaluating four variables.
  Flap Margin Assessment
  Papillae Evaluation
  Graft Site Examination
  Suture Evaluation
Modified Coronally advanced tunnel Difficulty score (MCATDS) for the treatment of gingival recessions | Baseline
  The MCATDS, developed by Górski in 2025 (Gorski et al. 2025), is a standardized scoring system to assess the complexity of treating multiple gingival recessions using the MCAT technique.
  The parameters include:
  * Tooth position (maxillary vs mandibular)
  * Tooth type (incisor/canine, premolar, molar)
  * Recession type (RT1, RT2, RT3)
  * Recession depth (<4 mm vs ≥4 mm)
  * Number of recessions involved (≤2, 3-4, ≥5)
  * Uniformity of recession sizes
  * Baseline keratinized tissue height
  * Gingival biotype (thick vs thin)
  * Frenulum presence and distance to gingival margin
  * Presence of scar tissue
  * Detectability of the cemento-enamel junction (CEJ)
  * Cervical step (>0.5 mm)
  * Tooth malposition
  Each parameter contributes between 0 and 2 points. The total score ranges from 0 to 17, and difficulty is categorized as:
  * Easy (0-5 points): Suitable for novice clinicians
  * Moderate (6-11 points): Requires experienced operators
  * Difficult (12-17 points): Reserved for highly skilled surgeons